CLINICAL TRIAL: NCT02320864
Title: A Pilot Study to Evaluate the Role of Brain Integrity on Post-hospital Sarcopenia
Brief Title: The Strong Brain Study
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201300566-N; P30AG028740 (NIH); 566-2013 (Other: UF legacy)
Record Dates: First submitted 2014-07-31; First posted 2014-12-19 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Osteoarthritis; Sarcopenia
Keywords: muscle strength; muscle weakness; hospitalization; surgery; total knee replacement
MeSH Terms: conditions — Osteoarthritis; Sarcopenia; Muscle Weakness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-surgical group: Adults who have knee osteoarthritis, but do not elect to have a total knee replacement surgery.
- Surgical group: Adults who have knee osteoarthritis and elect to have total knee replacement surgery.
  Interventions: Procedure: Total knee replacement surgery

INTERVENTIONS:
Procedure: Total knee replacement surgery — The surgeon removes damaged cartilage and bone from the surface of the knee joint and replaces them with a man-made surface of metal and plastic.
  Groups: Surgical group

SUMMARY:
To evaluate operational aspects of studying pre to post surgery/hospitalization changes in the integrity of a major white matter pathways and how these contribute to reductions in the ability to produce forceful muscle contractions.

DETAILED DESCRIPTION:
Hospitalization is a strong and independent risk factor for Sarcopenia. Older adults who are hospitalized in the previous year experience greater losses of lean mass and muscle strength than their non-hospitalized peers. Most of the research has focused on understanding muscle atrophy as the cause of weakness. However, post-hospitalization muscle weakness is not solely due to muscle atrophy- it explains less than 10% of the variance. The investigators propose that the sequela of hospitalization (e.g. deconditioning, disease severity, etc.) reduces the integrity of brain motor pattern that is used to produce forceful muscle contractions. Evidence from the literature suggests that central nervous system impairments explain approximately 60% of the variance in the loss in muscle strength observed following hospitalization. However, while these findings have helped to move the field forward, the measures lack spatial resolution. Accordingly, there remains a major gap in understanding whether deterioration of specific brain motor tracts contribute to post-hospitalization induced sarcopenia. The investigators intend to conduct a prospective cohort study to examine the integrity of the cortical-spinal white matter tract in post-hospitalized older adults. However, the investigators lack some essential elements in which to conduct this future study. Therefore, this pilot study will refine the following: patient eligibility, feasibility of collecting outcomes in patients, variances for statistical power, influence of covariates, timeline, patient attrition rates, data analysis strategies and magnetic resonance imaging protocol for mapping the cortical-spinal tract. The investigators will accomplish these operational aims efficiently and cost-effectively by leveraging funding with a newly awarded R01 by Dr. Catherine Price, which seeks to identify pre-surgical neuroimaging biomarkers following total knee arthroplasty (TKA) (R01NR014181; IRB# 487-2012). Specifically, the investigators will add measures of sarcopenia (muscle strength, mass and gait) and assess the integrity of the cortico-spinal tract. Measures will be collected in 20 patients before and after hospitalization (prior to surgery, 3 months and 12 months post-surgery) and 20 controls who are matched in age and disease severity at similar time points. In summary, there are long-term impairments that result from hospitalization in older adults that are not explained by the illness alone. This pilot study will result in subsequent larger NIH funded studies because the research is distinct from all others being conducted on muscle function, aging and effects of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years old or older with no upper limit at time of baseline assessment
* Right handed; restriction due to left-right hemisphere laterality and white matter pathways
* Able to understand and speak English
* Willing to give informed consent

Exclusion Criteria:

* Any conditions that pose health risk with physical exertion during a strength test as discovered on a medical history (e.g. heart failure, surgical complications etc.)
* Cancer requiring treatment in past 5 years (exception: non-melanoma skin cancer)
* Serious infectious diseases (e.g., self-reported HIV, sepsis)
* Myocardial infarction/ CVA within last six months
* Congestive heart failure (NY stage III or IV)
* Chronic hepatitis
* History of organ transplantation
* Seizure disorders
* History of head trauma resulting in intensive care
* Current diagnosis of alcoholism
* Drug dependence, or a history of major tranquilizer use
* History of major stroke(s)
* Exposure to toxins or neuroleptics
* History of encephalitis
* Neurological signs of upper motor neuron disease, cerebellar involvement, supranuclear palsy, or orthostatic hypertension that causes fainting
* Major Depression or Major Depressive Episode within three months prior to study
* Claustrophobia
* Non-medical bodily metal
* Pace-maker device
* Less than five years of formal education
* Inability to read or write
* Self-reported hearing or vision impairment that interferes with standardized test administration

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will comprise two age-matched participant groups: 1.) 'Healthy' non-demented (n=20) patients undergoing elective total knee arthroplasty, and 2.) age, education, and disease matched (osteoarthritis knee pain; n=20) non-surgery peers. We expect to screen 60 potential participants to yield 40 participants who complete the protocol. All participants will be recruited with the assistance of the Orthopedic Surgery Department at UFHealth. The parallel control group will originate from the parent study physician. Only right-handers will participate in this experiment because left-handedness is associated with greater variability in white matter organization and cognitive functions.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
muscle strength | Change in baseline, 3 months and 12 months
  We will measure plantar extension/flexion and knee extension/flexion strength using Isokinetic dynamometry (Biodex Inc., Shirley, NY). To prevent injury, participants will be secured to a padded chair using a lap and shoulder belts. To become accustomed to the testing machine, participants will first perform leg extensions with a light force applied to the target limb. Testing will commence after a short rest period that will be used to administer instruction and address any participant questions. Participants will perform 2 sets of each exercise for 15 repetitions at velocities of 60 degrees per second and 120 degrees per second. Tests will be done on both right and left sides and the maximal force will be determined. A 2-3 minute rest will be given between each set of exercise.
Muscle mass | Change in baseline, 3 months and 12 months
  Dual-energy X-ray absorptiometry (DEXA) whole body scan will be used to assess lean and fat mass of the lower extremity (Hologic, Discovery QDR Series, Bedford, MA). Participants will be asked to lie still on a table for approximately10 minutes while the scan is acquired by a certified technician.

SECONDARY OUTCOMES:
Short physical performance batter score (SPPB) | Change in baseline, 3 months and 12 months
  The SPPB test involves a brief performance battery based on timed short distance walk, repeated chair stands and balance test. Scores on each test is used to create a summary SPPB score that ranges from 0 (worst performers) to 12 (best performers).
6-minute walk distance | Change in baseline, 3 months and 12 months
  For the 6-minute walk test, participants will be asked to complete as much distance as possible on a circular walking course.
Spatiotemporal gait characteristics | Change in baseline, 3 months and 12 months
  step time, gait cycle, single support time, double support time, stance time, swing time, step length and stride length
Brain MRI derived corticospinal tract integrity from foot motor cortex to cerebral peduncle | Change in baseline, 3 months and 12 months
  This will be created by mapping two regions of interest: 1) Cerebral Peduncle and Foot/Left motor region. For the Cerebral Peduncle, we will use a method shown to be reliable (Triplett et al.). For the Foot/Left motor region, we will identify the foot cortex that will be guided by the areas of functional activation in the scanner and motor cortex regions of interest will be acquired from reliable raters.

OTHER OUTCOMES:
perceived pain | Change in baseline, 3 months and 12 months
  We will assess pain using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), and The Coping Strategies Questionnaire-Revised (CSQ-R). Pain ratings will also be collected during strength testing. Participants will be instructed to rate pain sensations experienced immediately prior, at mid-point during, immediately following, and 5 minutes post completion of the strength testing. Pain intensity will be measured on a scale of 0 (no pain sensation) to 100 (the most intense pain sensation imaginable).
physical activity | Change in baseline, 3 months and 12 months
  Participants will be asked to wear an accelerometer (Actigraph Inc, Pensacola, FL) that monitors physical movements (e.g. pedometer) on the waist following each testing session. The monitor will be placed around the waist using an elastic strap. They will be asked to wear the monitors for up to 10 days. Total physical activity time will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Todd M Manini, Ph.D., Principal Investigator — University of Florida; Adam J Woods, Ph.D., Principal Investigator — University of Florida
Locations (1):
- Institute on Aging, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided